CLINICAL TRIAL: NCT03651063
Title: Socially Assistive Robot in Upper-Limb Neurorehabilitation: A Long-Term Intervention RCT Using Behavioral Techniques
Brief Title: Socially Assistive Robot in Upper-Limb Neurorehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ben-Gurion University of the Negev (Other)
Responsible Party: Principal Investigator, Shelly Levy-Tzedek, Assistant Professor, Ben-Gurion University of the Negev
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5273-18-SMC
Record Dates: First submitted 2018-08-21; First posted 2018-08-29 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Upper Extremity Paralysis
Keywords: rehabilitation; social robots
MeSH Terms: interventions — Robotics

STUDY DESIGN:
Intervention Model Description: 3 groups, two groups each have a different intervention program, one control group with no intervention, only standard care.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- social robot group (Experimental)
  Interventions: Other: social robot
- computer group (Active Comparator)
  Interventions: Other: computer group
- contro: no intervention (No Intervention): This group will only be a follow up: clinical examination at the entrance and follow 5 weeks with clinical examination 5 weeks post, with no intervention.

INTERVENTIONS:
Other: social robot — Reach To Grasp games with a social robot
  Arms: social robot group
Other: computer group — reach to grasp games with a computer screen
  Arms: computer group

SUMMARY:
30 one year post stroke patients with upper limb paresis will be recruited to this study. The study is an RCT consists of two groups of intervention: 1. social robot, 2. computer, and one control group with no intervention. the intervention consists of 15 therapy sessions of reach-to-grasp games of the affected upper limb.

DETAILED DESCRIPTION:
Randomized Control Trial (RCT) longitudinal Intervention study. The RCT will be in accordance with the Consolidated Standards of Reporting Trials (CONSORT) statement . In this study there will be 2 groups of intervention and one control group:

1. Socially Assistive Robotic (SAR) intervention group.
2. Computer intervention group.
3. Control group: standard therapy. Participants A total of 30 subacute, one year post first stroke survivors, age 45-85, females and males, will be randomly allocated into 3 intervention groups. The participants will be recruited from Aleh Negev rehabilitation center, from the ambulatory day care by Dr. Oren Barzel-MD, a Rehabilitation Medicine specialist.

Procedure All patients that will be recruited to the study will be randomly allocated to each of the three intervention groups. The measurements and therapy sessions will take place in Aleh Negev rehabilitation center, in the Day-Care unit, by a physiotherapist and a PhD student from Ben Gurion University (GCP).

Evaluations for all patients will be conducted in three points of time: T1: entrance to the study, before randomization. T2: following 15 intervention sessions (after 5 weeks). T3: one month after end of the intervention. MMSE and FM-UE scores will be recorded as screening tools. FM-UE is a screening tool and a primary outcome measures. At each time point (T1, T2 and T3), the measurements described below will be performed on two separate days to avoid effect of fatigue. Participants will come for a total of 21 sessions: 2 sessions of evaluations, 15 sessions of treatment, 2 sessions of evaluation at the end of the intervention, 2 sessions of evaluations one month post intervention.

Intervention Program The intervention program consists of 15 therapy sessions, 3 times a week, an hour session each time for 5 weeks (over all 15 hours of intervention). Our proposed intervention is a graduated functional RTG games using real objects (like a cup or a jar), in different sizes, shapes, weights, textures and different environments (i.e. different heights or location on the table). The RTG game selected for a participant will be based on the upper limb movement and functional ability of the participant, as was measured by the therapist in the inclusion to the study. The progression will be starting from low table and progressing to higher table, starting from low weights objects (i.e. an empty jar) and progressing to higher weights (i. e. a jar full with flour). Our program is based on two critical parameters of upper limb rehabilitation: 1. the amount of practice-it has been recommended that individuals post-stroke perform as many repetitions per session as they can tolerate . 2. Practicing challenging tasks and not simple repetitive tasks, is likely to elicit motor learning and associated neural reorganization. Since a correlation between cognition and arm motor improvement has been lately described, the games we developed contain upper limb movement as well as cognitive aspects (like working memory). In each meeting the participant will have a one-hour session of RTG games, based on his\ her ability, as was measured upon enrollment in the study and based on his\her fatigue etc. The patient will be able to rest up to 5 minutes between a trial to trial in order to avoid fatigue. In addition, a patient will be able to stop a session at any time if desired. Even though our aim is to evaluate the motivation and performance of the patient outside the individual physiotherapy session with the therapist, we assume that during self-practice at the clinic and at home there is someone with the patient. Therefore during the therapy session of the intervention study a physiotherapist or a student will be present in the room (to help with problems that can arise). All sessions will be filmed and recorded upon agreement of the participant.

Group 1: Upper-limb functional RTG games with a humanoid robot (the "ROBOT group"). The robot that will be used in this study is the Pepper robot (Aldebaran Soft Bank robotics) -a humanoid off the shelf robot- with human-like face, 120 cm in height (see Figure 1). Pepper has a touch screen tablet on its chest. The participant will sit in front of the robot, and will play RTG games with the robot using real objects like a cup or a jar, open a drawer, order jars on a shelf etc. The robot will give the participant feedback on his\ her performance: the speed and the accuracy of the movement. There is no physical touch between the robot and he participant. There are no modulation of the off-the-shelf features of the robot for the study, besides recording the sentences of the robot speech for Hebrew in order for the patients to understand his speech. Pepper is off-the shelf humanoid robot, with human-like face. It can interact with the patient by gestures of voice (talk to the patient, encourage him\her to keep on training), by gestures of movement (like hand clapping, hand raising etc.) and by changing its color of eyes.

Group 2: Upper-limb functional RTG games with a computer (the "COMPUTER group"). The games are the same as described for the "ROBOT" group. In this group the pictures of the cups and the feedback on performance will be displayed on a standard computer screen (17''). There is no physical touch between computer and the participant.

Group 3: follow up with no intervention besides the usual rehabilitation program at the facility.

An example of a game: the cup game. In each trial, a row of colored cups will be displayed on the robot's chest tablet. The participant have to organize a corresponding set of actual physical cups on the table according to the picture shown on the screen. There are three levels of game difficulty: in Level 1 participants are asked to arrange four cups in the correct order, in Level 2 there are five cups, and in Level 3 there are six cups. The instructions and feedback will be provided by either the robot, or displayed on the computer screen or written on a paper. The picture with the target order of the cups will disappear from the screen after 1-2 min. In the computer and robot groups, when they complete the task, participants will have to press a push button. In the robot and computer groups, after each trial, the robot\ computer will either give feedback on the performance (e.g., "try to do it faster next time") or a feedback on results (e.g., "you succeeded!", "you were not right but try again!"). The feedback given by the robot is both verbal and with head and arm gestures (e.g. hand clapping). The feedback by the computer will be displayed on the screen. In the self-training group no feedback is given. After two trials on the basic level (four cups) and four trials on the second level (five cups), the participant could choose to either continue at the same level or change to a harder level of game (more cups).

A. Games description and progression

1. The cup game: Ordering a row of cups according to the picture. Progression 1: number of cups: start from 3 cups, continue to 6 cups. Progression 2: Height of table: start low, continue to high, continue to different heights, different weights of cups.
2. A dartboard: ordering cups on a dartboard according to a picture. Progression 1: number of cups: start from 3 cups continue up to 7 cups.

   Progression 2: start close to body (at arm's length) continue longer than arm length. Progression 3: height of table. Progression 4: weight of cups.
3. Ordering Jars on different heights shelves: according to a picture. Progression 1: start 3 jars, add jars. Progression 2: start low height, continue high and different heights. Progression 3: different weights of jars.
4. Open drawer and order objects according to a picture (memory game). Progression 1: number of drawers-start with 2 and add drawers. Progression 2: different heights drawers. Progression 3: start with a handle of different kinds (straight handle, round handle) continue to a key opening.
5. Taking objects (i.e. keys) out of a jar and putting it in a jar according to its color (stroop game).

ELIGIBILITY:
Inclusion Criteria:

1. First unilateral stroke (ischemic or hemorrhagic)
2. Mini-Mental State Examination (MMSE) score ≥ 24/30
3. Fugl-Meyer Upper Extremity (FM-UE) score 16-66
4. Upper limb muscle tone assessed by Modified Ashworth Scale ≤ 2
5. Ability of the participant to sit independently without external support. -

Exclusion Criteria:

1. Additional neurological or musculoskeletal problems (such as Parkinson's disease, unilateral neglect, Pusher syndrome and apraxia).
2. Severe vision or sensory deficits affecting upper limb movements.
3. Aphasia affecting understanding of simple instructions.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Sensory Motor Recovery of the upper limb | 20 minutes
  upper limb impairment assessment will be assessed by the Fugl-Meyer Assessment. This is the gold-standard assessment for upper limb motor ability in stroke patients. It comprises of 33 items.
The amount of use of the upper extremity in everyday life | 15 minutes
  The Motor Activity Log: a questionnaire consist of items regarding the use of the affected arm in every day tasks

SECONDARY OUTCOMES:
index of curvature | 30 minutes
  The ratio between a straight line and the path of the movement the participant did.
stroke impact scale | 30 minutes
  questionnaire regarding the effect of stroke on different aspects of life such as motor, cognitive, emotional and communication

OTHER OUTCOMES:
Perceived Competence (Exercising Regularly) questionnaire | 5 minutes
  4 items scale regarding the motivation of a person to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Shelly Levy-Tzedek, PhD, Study Chair — Ben-Gurion University of the Negev
Locations (1):
- Aleh Negev Rehabilitation Center, Ofakim, South, Israel

REFERENCES:
- [Derived] Feingold-Polak R, Barzel O, Levy-Tzedek S. Socially Assistive Robot for Stroke Rehabilitation: A Long-Term in-the-Wild Pilot Randomized Controlled Trial. IEEE Trans Neural Syst Rehabil Eng. 2024;32:1616-1626. doi: 10.1109/TNSRE.2024.3387320. Epub 2024 Apr 19. PMID 38598401
- [Derived] Feingold-Polak R, Barzel O, Levy-Tzedek S. A robot goes to rehab: a novel gamified system for long-term stroke rehabilitation using a socially assistive robot-methodology and usability testing. J Neuroeng Rehabil. 2021 Jul 28;18(1):122. doi: 10.1186/s12984-021-00915-2. PMID 34321035